CLINICAL TRIAL: NCT06249919
Title: A Phase 1b/2a, Double-blinded, Placebo-controlled, Multiple Doses, 2 Step-up Study Evaluating the Safety, Tolerability, PK/PD and Efficacy of Systemic NS101 in Healthy Volunteers and SSNHL Patients
Brief Title: A Phase 1b/2a, Study Evaluating the Safety, PK/PD and Efficacy of NS101 in Healthy Volunteers and SSNHL Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Neuracle Science Co., LTD. (Industry)
Collaborators: Samsung Medical Center (Other); Severance Hospital (Other); Korea University Anam Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NS101_P2_04
Record Dates: First submitted 2024-01-12; First posted 2024-02-08 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Seneorineural Deafness; Sudden Sensorineural Hearing Loss
Keywords: Sensorineural disease; sudden sensorineural hearing loss; sensorineural hearing loss; sudden deafness; cochlear synaptopathy; hidden auditory synaptopathy
MeSH Terms: conditions — Hearing Loss, Sudden; Hearing Loss, Sensorineural; Hearing Loss, Hidden

STUDY DESIGN:
Intervention Model Description: A Phase 1b/2a, prospective, randomized, double-blind, placebo-controlled, multicenter, dose-escalation, exploratory study evaluating the safety, tolerability, pharmacokinetics/pharmacodynamics (PK/PD), and efficacy of multiple doses of NS101 in healthy adults and patients with sudden Sensorineural Hearing Loss
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group A (Experimental): NS101 15mg/kg IV infusion Biweekly for 6weeks in Healthy Volunteers (active:placebo=6:3)
  Interventions: Biological: NS101; Biological: Placebo
- Group B (Experimental): NS101 30mg/kg IV infusion Biweekly for 6weeks in Healthy Volunteers (active:placebo=6:3)
  Interventions: Biological: NS101; Biological: Placebo
- Cohort A (Active Comparator): NS101 15mg/kg IV infusion Biweekly for 12weeks in Sudden Sensorineural Hearing Loss patients
  Interventions: Biological: NS101
- Cohort B (Placebo Comparator): Placebo 15mg/kg IV infusion Biweekly for 12weeks in Sudden Sensorineural Hearing Loss patients
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: NS101 — NS101 is anti FAM19A5 antibody expected to play as a synapse organizer and reversing synapse dysfunction in various neurological diseases
  Arms: Cohort A; Group A; Group B
Biological: Placebo — Placebo (i.e. fake drug without active pharmaceutical ingredient) of NS101
  Arms: Cohort B; Group A; Group B

SUMMARY:
The goal of this 2 step-up, exploratory study is to test safey, tolerability and PK/PD profiles in healthy volunteers and safety, tolerability and efficacy in sudden sensorineural hearing loss patients as an early salvage therapy.

The main questions it aims to answer are:

1. whether is it safe and tolerable when healthy volunteers and sudden sensorineural hearing loss patients take multiple doses of NS101 against FAM19A5
2. whether is it effective in reversing hearing capability in sudden sensorineural hearing loss patients who fails to show sufficient recovery despite of oral standard steroid therapy.

Patients and heathly volunteers will be given NS101 15mg/kg or 30mg/kg systemically less than 3 months per protocol.

This is placebo controlled, double blinded study, which means there will be a group who receives placebo (i.e. fake drug) for study purpose.

ELIGIBILITY:
Part A: healthy volunteers

Part B:

Inclusion Criteria:

* unilateral ideopathic SSNHL greater than 45dB at the average of 4 frequencies in PTA (contralateral hearing is less than 30dB)
* Subject who has completed investigator-recognized standard treatment within 30 days of symptom onset and is able to undergo randomization visit within 35 days.
* Subjects who, in the opinion of the investigator, have received sufficient systemic steroid therapy for approximately 2 weeks recovery
* A combination regimen consisting of approximately 2 weeks of systemic steroid therapy and intratympanic steroid administration

Exclusion Criteria:

* other otologic or systemic diseases
* retrocochlear lesion

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1b part: Change from Baseline in Safety Profiles | Baseline, Day1, Day2, Day3, Day14, Day15, Day16, Day17, Day28, Day29, Day30, Day32, Day43
  Adverse Event, Serious Adverse Event, ratio of Treatment related Serisous Adverse Event with causality & severity will be descriptively measured and collected in the following time frames
Phase 2a part: Changes from Baseline in Safety Profiles | Baseline, Week1, Week2, Week4, Week6, Week8, Week10, Week12, Week16, Week20
  Adverse Event, Serious Adverse Event, ratio of Treatment related Serisous Adverse Event with causality & severity will be descriptively measured and collected in the following time frames

SECONDARY OUTCOMES:
Phase 1b part: Change from Baseline in PK/PD profiles & Immunological Assay | Baseline, Day1, Day2, Day3, Day14, Day15, Day16, Day17, Day28, Day29, Day30, Day32, Day43
  Concentrations, Areas Under the Curve versus time curve, Times and Volumes of Distribution of various status verus time curve
Phase 2a part : Change from Baseline in PK/PD profiles & immunological Assay | Baseline, Week1, Week2, Week4, Week6, Week8, Week10, Week12, Week16, Week20
  Concentrations, Areas Under the Curve versus time curve, Times and Volumes of Distribution of various status verus time curve

OTHER OUTCOMES:
Phase 2a part : Change from Baseline in Pure Tone Audiometry, Speech Discrimination Scores and Tinnitus Handicap Inventory in Sudden Sensorineural Hearing Loss Patients | Baseline, Week4, Week8, Week12, Week16, Week20
  hearing capacity of thresholds (e.g. PTA, ABR, DPOAE, ECochG), speech discrimination (e.g. SRT, SDS) and tinnitus (e.g. THI, VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Park, M.D., Study Director — Neuracle Science
Locations (15):
- South Korea (15):
  - SCH University Hospital Bucheon, Bucheon-si
  - Chonam National University Hospital, Gwangju
  - Inje University Ilsan Paik Hospital, Ilsan
  - Myongji Hospital, Ilsan
  - Pusan National University Hospital, Pusan
  - Hallym Sacred Heart Hospital, Pyeongchon
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Catholic University Seoul St. Mary's Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Yonsei University Severance Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: No
Currently there is no plan to share IPD at this stage